CLINICAL TRIAL: NCT03040635
Title: An Investigator/Subject Blind, Randomized, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of RO7034067 in Healthy Japanese Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Risdiplam (RO7034067) in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP39625
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Risdiplam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Risdiplam '2' Milligrams (mg) (Experimental): A single dose of 2 mg Risdiplam will be administered to all participants randomized to this arm under fasted conditions as an oral drinking solution on Day 1.
  Interventions: Drug: Risdiplam
- Risdiplam '6' mg (Experimental): A single dose of 6 mg Risdiplam will be administered to all participants randomized to this arm under fasted conditions as an oral drinking solution on Day 1.
  Interventions: Drug: Risdiplam
- Risdiplam '12' mg (Experimental): A single dose of 12 mg Risdiplam will be administered to all participants randomized to this arm under fasted conditions as an oral drinking solution on Day 1.
  Interventions: Drug: Risdiplam
- Placebo (Placebo Comparator): A single dose of placebo will be administered to all participants randomized to this arm under fasted conditions as an oral drinking solution on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risdiplam — Single oral doses of Risdiplam will be administered on Day 1.
  Other Names: RO7034067
  Arms: Risdiplam '12' mg; Risdiplam '2' Milligrams (mg); Risdiplam '6' mg
Drug: Placebo — Single oral doses of Risdiplam matching placebo will be administered on Day 1.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single oral doses of Risdiplam in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants of Japanese origin, with Japanese parents (for the provisional Caucasian cohort, participants must be male or female Caucasians with 4 Caucasian grand-parents)
* Healthy participants. Healthy status is defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including ophthalmological examination, vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* A body mass index (BMI) between 18 to 30 kilograms per square meter (kg/m^2) inclusive
* Male participants must agree to use a barrier method of contraception from dosing until completion of the study and for 4 months thereafter
* Female participants must be either surgically sterile or post-menopausal

Exclusion Criteria:

* Medical history of cardiovascular disease, renal disease, liver disease, digestive system disease, blood dyscrasia, immunologic disease, diseases of the nervous system, endocrine disease, metabolic disease, lung disease, or with anamnesis and obstacles in kidney, liver, or cardiopulmonary function
* Participants with any clinically significant eye pathology
* Laboratory test (hematology, biochemistry, physical examination or vital signs) values outside the institutional normal range and rated as clinically significant abnormal at screening
* Any clinically significant abnormalities in ECG at screening
* Inherited long QT syndrome or known family history of arrhythmia
* Systolic blood pressure (SBP) higher than 140 millimeters of mercury (mmHg) or below 90 mmHg, and/or diastolic blood pressure (DBP) higher than 90 mmHg or below 50 mmHg in the supine position, as assessed at screening
* Positive result for human immunodeficiency virus (HIV) antigen and antibody, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody at screening
* Donation or loss of blood over 500 milliliters (mL) within three months prior to screening
* History of smoking more than 10 cigarettes a day. Participants who have quit smoking or who have reduced their daily cigarette smoking to 10 or less for more than one month prior to screening are allowed
* Daily consumption of food or drink containing a large amount of methylxanthine (caffeine, theophylline, theobromine)
* Present or past history of substance addiction, dependence or abuse, such as abuse of drugs or alcohol
* Concomitant or previous participation in any clinical trial either within 90 days or 5 half-lives of the investigational drug, whichever is longer, before administration of study drug in this study
* Use of prescribed medications which have systemic exposure within one week before enrolment
* Use of any concomitant drug during the study (including over-the-counter medication and medications used in dentistry)
* Inability to meet the study requirements in the opinion of the Investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Risdiplam | Pre-dose (0 hour [hr]), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Time to Maximum Plasma Concentration (Tmax) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Area Under the Plasma Concentration-Time Curve up to the Last Measurable Concentration (AUClast) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Area Under the Plasma Concentration-Time Curve up to Time t (AUC0-t) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Apparent Terminal Half-Life (t1/2) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Apparent Oral Clearance (CL/F) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Apparent Oral Volume of Distribution (Vz/F) of Risdiplam | Pre-dose (0 hr), 0.5, 1, 2, 3, 4, 4.5, 5, 6, 8, 10, 12, 24, 36, 48, 72, 120, 168, 264 hr postdose from Day 1
Cumulative Amount Excreted Unchanged into Urine (Ae) of Risdiplam | Pre-dose (0 hr), and 5 urine samples at different time-ranges postdose (0-6 hr, 6-12 hr, 12-24 hr, 24-48 hr, and 48-72 hr)
Renal Clearance (CLR) of Risdiplam | Pre-dose (0 hr), and 5 urine samples at different time-ranges postdose (0-6 hr, 6-12 hr, 12-24 hr, 24-48 hr, and 48-72 hr)
Fraction of Dose Excreted Unchanged Renally (Fe) of Risdiplam | Pre-dose (0 hr), and 5 urine samples at different time-ranges postdose (0-6 hr, 6-12 hr, 12-24 hr, 24-48 hr, and 48-72 hr)
Percentage of Participants with Adverse Events (AEs) | Up to approximately 7 weeks

SECONDARY OUTCOMES:
Change from Baseline in Splicing Modifications of Survival of Motor Neuron (SMN) Messenger Ribonucleic Acids (mRNAs), Including SMN1, SMN2 Full Length (FL), and SMNdelta7 mRNA in Blood In Vivo | Days -1, 1, 2, 3, 4, 6
Change from Baseline in mRNA Levels of Paired Box (PAX) Genes in Blood | Days -1, 1, 2, 3, 4, 6
Change from Baseline in SMN Protein Levels in Blood | Day -1, follow-up visit (Day 21)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Collaborative Neuroscience Network, Inc., Garden Grove, California, United States

IPD SHARING:
Plan to Share IPD: Undecided